CLINICAL TRIAL: NCT00653835
Title: SCH 58235: A Multicenter, Randomised, Parallel Groups, Placebo-Controlled Study Comparing The Efficacy, Safety, and Tolerability Of The Daily Co-Administration of Ezetimibe 10 mg With Simvastatin 20 mg vs Ezetimibe Placebo With Simvastatin 20 mg in Untreated Subjects With Primary Hypercholesterolaemia And Coronary Heart Disease (Protocol P03435)
Brief Title: Ezetimibe Plus Simvastatin Versus Simvastatin in Untreated Subjects With High Cholesterol (P03435)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P03435
Record Dates: First submitted 2008-04-01; First posted 2008-04-07 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolaemia; Atherosclerosis
MeSH Terms: conditions — Hypercholesterolemia; Atherosclerosis | interventions — Ezetimibe, Simvastatin Drug Combination; Ezetimibe; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Ezetimibe + Simvastatin (Experimental)
  Interventions: Drug: Ezetimibe + Simvastatin
- Simvastatin (Active Comparator)
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Ezetimibe + Simvastatin — oral tablets: ezetimibe 10 mg + simvastatin 20 mg once daily for 6 weeks
  Other Names: SCH 58235; Zetia; Zocor
  Arms: Ezetimibe + Simvastatin
Drug: Simvastatin — oral tablets: simvastatin 20 mg + ezetimibe placebo once daily for 6 weeks
  Other Names: Zocor
  Arms: Simvastatin

SUMMARY:
This study will assess whether co-administration of ezetimibe 10 mg with simvastatin 20 mg will be more effective than treatment with simvastatin 20 mg alone in reducing LDL-C concentrations when administered for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years and <= 75 years of age
* LDL-C concentration >= 3.3 mmol/L (130 mg/dL) to <= 4.9 mmol/L (190 mg/dL) at baseline.
* Triglyceride concentration <3.99 mmol/L (350 mg/dL) at baseline.
* Documented coronary heart disease (CHD), which will include one or more of the following features: documented stable angina (with evidence of ischemia on exercise testing); history of MI; history of PCI (primarily PTCA with or without stent replacement); symptomatic peripheral vascular disease; documented history of atherothrombotic cerebrovascular disease; and/or documented history of non-Q wave MI.
* Stable weight history for at least 4 weeks prior to entry into study at baseline.
* Female subjects of childbearing potential must be using an acceptable method of birth control or be surgically sterilized.

Exclusion Criteria:

* Body mass index (BMI) >=35 kg/m^2 at baseline.
* Subjects whose liver transaminases (ALT, AST) are >1.5 times the upper limit of normal and with active liver diseases at baseline.
* Subjects with evidence of current myopathy (including subjects with CK>1.5 times above the upper limit of normal) at baseline.
* Subjects with clinical laboratory tests (CBC, blood chemistries, urinalysis) outside the normal range that are clinically acceptable to the investigator at baseline.
* Subjects with Type II diabetes mellitus who are poorly controlled (HbA1c>9%) or newly diagnosed (within 3 months) or who have had a change in anti-diabetic therapy within 3 months of baseline.
* Subjects with Type I diabetes mellitus who have not been on a stable insulin regimen for 3 months prior to baseline, or who have a recent history of repeated hypoglycaemia or unstable glycaemic control.
* Subjects who have known hypersensitivity to HMG-CoA reductase inhibitors.
* Female subjects who consume >14 units and male subjects who consume >21 units of alcohol per week.
* Female subjects who are pregnant or breast feeding.
* Subjects who have not observed the designated washout periods for any of the prohibited medications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2003-09-01 (Actual); Primary Completion 2004-08-01 (Actual); Study Completion 2004-08-01 (Actual)

PRIMARY OUTCOMES:
Percent change in LDL-C from baseline to endpoint. | 6 weeks

SECONDARY OUTCOMES:
Percent of subjects who achieve LDL-C ESC goal (ie, <3 mmol/L [115 mg/dL]) at endpoint. | 6 weeks
Percent change from baseline to endpoint in total cholesterol, HDL-C and triglycerides. | 6 weeks
Safety: adverse events, laboratory test results, vital signs. | Throughout study

REFERENCES:
- [Result] Patel JV, Hughes EA. Efficacy, safety and LDL-C goal attainment of ezetimibe 10 mg-simvastatin 20 mg vs. placebo-simvastatin 20 mg in UK-based adults with coronary heart disease and hypercholesterolaemia. Int J Clin Pract. 2006 Aug;60(8):914-21. doi: 10.1111/j.1742-1241.2006.01023.x. PMID 16893434